CLINICAL TRIAL: NCT03726905
Title: Effectiveness and Safety of Complex Exercises of the Respiratory Muscles Plus Aerobic Training vs. Aerobic Training in Patients With CHF and II-IV NYHA FC: Prospective Randomized Clinical Trial With Sham Control
Brief Title: Complex Exercises of the Respiratory Muscles Plus Aerobic Training vs. Aerobic Training in Patients With СHF
Acronym: AEROFIT-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lomonosov Moscow State University Medical Research and Educational Center (Other)
Collaborators: Russian Heart Failure Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mcmsuaadd001
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure
Keywords: CHF; exercise; aerobic; respiratory muscle training
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: The control group will be assigned an imitation of respiratory muscles training with the help of breathing simulators, with a breathing resistance level set at 0
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- respiratory muscles training (Experimental): 4 weeks guided respiratory muscles training followed by 12 weeks guided aerobic training - (treadmill walking)
  Interventions: Other: respiratory muscles training; Other: aerobic training
- sham respiratory muscles training (Sham Comparator): 4 weeks sham respiratory muscles training (THRESHOLD® IMT breathing trainer with "0" pressure level) followed by 12 weeks guided aerobic training - (treadmill walking)
  Interventions: Other: sham respiratory muscles training; Other: aerobic training

INTERVENTIONS:
Other: respiratory muscles training — 4 weeks respiratory muscles training aimed on respiratory muscles endurance and lengthening expiration time
  Arms: respiratory muscles training
Other: sham respiratory muscles training — 4 weeks sham respiratory muscles training with the help of breathing simulators, with a breathing resistance level set at 0
  Arms: sham respiratory muscles training
Other: aerobic training — 12 weeks treadmill walking

SUMMARY:
The aim of the study is to test the hypothesis that the physical rehabilitation starting with respiratory training followed by the aerobic exercises will have a more pronounced effect on clinical and functional indicators than the currently used physical rehabilitation based on aerobic training alone

DETAILED DESCRIPTION:
Changes in the respiratory muscles play an important role in the pathophysiology of exercise intolerance in CHF patients. The weakness of the respiratory muscles leads to a decrease in the efficiency of breathing and the formation of a pathological type of breathing, in which the inhalation time is prolonged, and the expiration time is shortened. Patients with weak respiratory muscles have impaired functional status, as determined by peak oxygen consumption. The violation of the ratio of inspiratory time / to the total time of the respiratory cycle is associated with an increase in the activity of the sympathoadrenal system. The positive effect of respiratory muscle training on MIP, MEP, peak VО 2, VE, VE / VCO 2 slope, VE oscillation, rhythm variability, and quality of life parameters is shown. Decreased oxygenation of the respiratory muscles during intense physical exertion in patients with CHF may increase respiratory failure and provoke hyperactivation of the inspiratory metaboreflex, thereby aggravating exercise intolerance due to a decrease in muscular-muscular system perfusion due to redistribution of blood flow. In addition, it was shown that fatigue of the respiratory muscles increases the activity of the sympathetic nervous system and reduces blood flow in the muscles of the inactive limb due to adrenergic vasoconstriction. This response is most likely associated with metabolic stimulation of small afferent type III and IV fibers of the respiratory muscles, especially the diaphragm. Respiratory muscle training can minimize the effects of inspiration metaboreflex activation and prolong the duration of exercise. In addition, several studies have shown that the strength of the respiratory muscles in patients with HF correlates with central hemodynamic indices at rest, including cardiac output, mean pulmonary pressure and pulmonary vascular resistance. Several studies have shown that the mechanism that improves exercise tolerance in patients with HF after training the respiratory muscles is to increase the blood supply to the muscles of the limbs at rest and during exercise. Thus, the mechanisms of the effect of the weakness of the respiratory muscles on the pathogenesis of a decrease in the functional ability of patients are well studied. Both respiratory muscular and aerobic exercises of moderate effectiveness are recommended by leading medical communities as an effective means to improve the functional ability of patients, improve quality of life parameters, improve symptoms and reduce hospital admissions (level of evidence Level 1). At the same time, respiratory muscle training is recommended as the beginning of physical rehabilitation in patients with IV FC HF, and moderate-intensity aerobic training is recommended for patients with FC I-III FC. Also, in individual works abroad, the effects of respiratory muscle training on clinical CHF. However, according to the investigator's information, no studies have been carried out on the study of the method of functional training, including training of the respiratory muscles, as an obligatory initial stage of physical rehabilitation of patients with any functional class of HF.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years and older (inclusive)
* Patients with stable heart failure of the II-III functional class.
* Signed patient informed consent to participate in the study.
* Left ventricular ejection fraction ≤40%, confirmed by the results of EchoCG no more than 3 months before the start of the study.
* Patients who can understand the objectives of this study and comply with the requirements of the Protocol.

Exclusion Criteria:

* • Heart failure I and VI functional class

  * Left ventricular ejection fraction> 41% or no confirmed data on the left ventricular EF.
  * Myocardial infarction, ACS, heart surgery, percutaneous coronary intervention, or coronary artery bypass surgery performed less than 3 months prior to randomization.
  * Unstable or refractory angina.
  * Pulmonary heart.
  * Constrictive pericarditis.
  * Hypertrophic cardiomyopathy.
  * Amyloid cardiomyopathy.
  * Syndrome of premature excitation of the ventricles.
  * The need for percutaneous coronary intervention or coronary bypass surgery in the near future.
  * Sinus node dysfunction syndrome.
  * The presence of a pacemaker.
  * The presence of diagnosed non-cardiac causes of CHF.
  * Any non-cardiac disease that reduces the expected duration to less than 2 years from the moment of randomization.
  * A stroke less than 1 month prior to randomization or a stroke with marked continuing neurological disorders less than 12 months before randomization
  * Orthopedic disorders that prevent physical training
  * COPD, Bronchial asthma. Another lung disease that can affect CSTP results
  * Significant impaired renal function (plasma creatinine 220 µmol / L or higher).
  * Significant abnormal liver function (increased ALT or AST more than 3 times relative to the upper limit of normal).
  * Acute coronary syndrome less than 3 months before randomization.
  * Obstructive or restrictive cardiomyopathy.
  * Acute myocarditis.
  * Hemodynamically significant organic lesions of valves requiring surgical intervention.
  * A history of heart transplantation or current waiting for a heart transplant.
  * Drug addiction, substance abuse, alcoholism, drug use in history.
  * Mental, physical and other reasons that do not allow to adequately assess their behavior and correctly fulfill the conditions of the study protocol.
  * A history of any significant, in the opinion of the physician-researcher, condition / disease or circumstances that prevent the inclusion in the study.
  * Inability / reluctance of the patient to provide signed informed consent to participate in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Functional Capacity | 16 weeks
  Change in Peak VO2

SECONDARY OUTCOMES:
proBNP | 4 weeks
  Change in concentration of NT- proBNP from baseline
proBNP | 16 weeks
  Change in concentration of NT- proBNP from baseline
Respiratory muscle strength | 4 weeks
  Change in maximal inspiratory and expiratory pressures (PImax and PEmax) from baseline
Respiratory muscle strength | 16 weeks
  Change in maximal inspiratory and expiratory pressures (PImax and PEmax) from baseline
Neurohormone activity | 4 weeks
  Difference between Active and Control groups in Angiotensin II (A II) concentration from baseline
Neurohormone activity | 16 weeks
  Change in concentration of Angiotensin II (A II) from baseline

OTHER OUTCOMES:
Change in health-related quality of life | 4 weeks
  Minnesota Living with Heart Failure Questionnaire/ The quality of life between study groups and the change in quality of life over time between study groups.
Change in health-related quality of life | 16 weeks
  Minnesota Living with Heart Failure Questionnaire. Assessed from baseline visit to 16 weeks follow-up visit.The quality of life between study groups and the change in quality of life over time between study groups using clinically accepted quality of life measures. MLHFQ
Anxiety and Depression | 4 weeks
  Hospital Anxiety sand Depression Scale (HADS) The questionnaire comprises seven questions for anxiety and seven questions for depression.Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21. The cut off for both scales in 11.
Anxiety and Depression | 16 weeks
  Hospital Anxiety sand Depression Scale (HADS) The questionnaire comprises seven questions for anxiety and seven questions for depression.Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21. The cut off for both scales in 11.

CONTACTS AND LOCATIONS:
Overall Officials: Yana A Orlova, Professor, Study Chair — Moscow State University
Locations (1):
- Julia Begrambekova, Moscow, Moscow Oblast, Russia

IPD SHARING:
Plan to Share IPD: No